CLINICAL TRIAL: NCT06165419
Title: A Phase II Study Evaluating Definitive Radiosurgical Decompression in Patients With High-Risk Spinal Metastases
Brief Title: Definitive Radiation for High-Risk Spine Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kartik Mani, Assistant Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBU-RT-MESCC; IRB2023-00421 (Other: Stony Brook University)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Cancer; Metastatic Lung Cancer; Metastatic Breast Cancer; Metastatic Tumor; Metastatic Tumor of Bone; Metastatic Tumor to the Spine; Spine Metastases; Metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SBRT to the spine (Experimental)
  Interventions: Radiation: SBRT to the spine

INTERVENTIONS:
Radiation: SBRT to the spine — Stereotactic body radiation therapy (SBRT) administered to spine metastases

SUMMARY:
This study is looking at whether patients with cancer that has aggressively spread to the spine can be treated with stereotactic body radiation therapy only and avoid a large spine surgery

ELIGIBILITY:
Eligible patients must have:

* Any pathologically proven solid tumor diagnosis not of central nervous system origin with radiographic or pathologic evidence of metastatic disease
* Metastatic spine involvement documented by imaging
* Involvement of maximum 3 contiguous vertebral bodies at the index site
* Intact neurologic function, or only minor neurologic deficits with muscle strength greater or equal to 4 out of 5 with or without steroids
* An evaluation by an radiation oncology and orthopedic spine/neurosurgery attending
* ECOG Performance Status of 0-3

Patients are ineligible if they have:

* An unstable spine defined as a Spinal Instability Neoplastic Score (SINS) greater than 12
* Had previous surgery or radiation to address the target spinal metastases
* Radiosensitive tumors (e.g. small cell lung cancer, lymphoma, multiple myeloma, and germ-cell tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of spinal surgery/stabilization within 6 months following SBRT | 6 months
  Assess the efficacy of spine SBRT alone in controlling spine metastases

SECONDARY OUTCOMES:
Reduction in epidural tumor volume | 3 months
  Percent reduction of epidural volume of the treated metastatic lesions
Changes on Neck Disability index | 1 months, 3 months, 6 months
  The Neck Disability Index measures neck pain and disabilities in patients with neck pain, with scores varying from 0 to 50. Lower scores indicate better outcomes, higher scores indicate a worse outcome.
Changes on Oswestry Low Back Disability Questionnaire | 1 months, 3 months, 6 months
  The Oswestry Disability Index measures disability in patients with low back pain, with scores varying from 0 to 50. Lower scores indicate better outcomes, higher scores indicate a worse outcome.
Changes on EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire | 1 months, 3 months, 6 months
  The EuroQol 5D-5L questionnaire measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each health dimension is scored from 1 to 5, with 1 indicating a better health state, and 5 the worse state possible. Respondents also indicate their overall health status on visual analogue score, with values ranging from 0 (worst health imaginable) to 100 (best health imaginable)
Progression-free survival | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Mani, MD PhD, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No